CLINICAL TRIAL: NCT00695916
Title: Randomized Trial of Breast MRI in Women With Newly Diagnosed Breast Cancer Prior to Breast Conserving Surgery
Brief Title: MRI in Women With Newly Diagnosed Breast Cancer Prior to Breast Conserving Surgery
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: PI
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BRSNSTU0025; 98272 (Other: Stanford University Alternate IRB Approval Number); BRSNSTU0025 (Other: [Stanford University OnCore Number); NCT00695916 (Other: ClinicalTrails.gov); 6125 (Other: Stanford IRB)
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Procedure: Breast MRI

SUMMARY:
To see if performing breast MRI before a lumpectomy will help the surgeon successfully remove the entire cancer with normal tissue margins in a single operation thereby reducing the need for additional surgical procedures. The study will also measure how well MRI can find unsuspected cancers in the same breast as the known cancer; how well MRI will find unsuspected cancers in the opposite breast; how often MRI will generate false positive MRI findings; whether routinely incorporating breast MRI delays care or adds unnecessary cost; and, whether breast MRI is able to reduce the frequency of cancer recurrence in the treated breast or elsewhere in the body.

ELIGIBILITY:
Inclusion Criteria:

* DCIS less than 5 cm. T1/T2 invasive breast cancer. Patient is a suitable candidate for breast conservation and wishes this as the primary clinical approach
* No breast MRI within the past year. Prior core biopsy, but no prior excision allowed. Patient has completed conventional imaging workup with mammography ultrasound as indicated and there is no clinical indication for breast MRI.
* Women with age >= 18. No ethnic restrictions.
* No life expectancy restrictions.
* Performance status not a factor.
* No requirements for organ or marrow function.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patient is unable to complete a breast MRI due to such factors as hardware and claustrophobia.
* No limitations as to other investigational agents. Patients who have received neoadjuvant chemotherapy will not be included in the study due to the limitations of MRI interpretation after neoadjuvant chemotherapy and because this represents a distinct scenario for interpretation of breast MRI in comparison with untreated patients.
* There are no comorbidities that would preclude entry into the study unless the patient is unable to lay still for breast MRI scanning.
* There are fewer reactions to MRI contrast media, but if there is such a history, the patient will be excluded from consideration.
* There are no exclusion criteria based on concomitant medications.
* There are no other agent specific exclusion criteria.
* Pregnancy is considered a contraindication given the uncertain effects of breast MRI on the fetus.
* Cancer survivors are candidates for the study unless the patient has a prior ipsilateral breast tumor.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To determine whether pre-lumpectomy breast MRI reduces the frequency of repeat lumpectomy in women with DCIS < 5 cm or T1 or T2 invasive breast cancer

SECONDARY OUTCOMES:
To determine how often MRI will detect occult multifocal or multicentric disease
To determine how often MRI will miss occult DCIS or invasive cancer subsequently detected on surgical pathology
To determine the frequency with which breast MRI changes the surgical plan
To determine the frequency of false positive MRI findings requiring biopsy
To measure whether MRI reduces the frequency of repeat lumpectomy to a greater extent in women with mammographically dense vs fatty breasts
To measure whether preoperative MRI is associated with enhanced postoperative cosmesis
To measure whether preoperative MRI alters cost of care
To measure the degree and extent to which preoperative MRI lengthens the time required to deliver care
To measure whether preoperative MRI increases the rate of patient directed ("unnecessary") mastectomy
To measure whether MRI decreases the risk of ipsilateral breast tumor recurrence
To measure disease-free survival without/with preoperative breast MRI
To measure overall survival without/with preoperative MRI

CONTACTS AND LOCATIONS:
Overall Officials: Frederick M. Dirbas, Principal Investigator — Stanford University